CLINICAL TRIAL: NCT06264076
Title: Ligament Balancing in Total Knee Arthroplasty - A Proof-of-Concept Study on a Systematic Approach to Bellemans Technique
Brief Title: Ligament Balancing in Total Knee Arthroplasty
Acronym: BLIS-TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Lars Engseth, MD, orthopaedic consultant, Oslo University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 686340; CIV-NO-23-09-043976 (Other: Eudamed CIV ID)
Record Dates: First submitted 2024-02-01; First posted 2024-02-16 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Ligament; Laxity, Knee; Knee Osteoarthritis
Keywords: Total knee arthroplasty (TKA); Total Knee Replacement (TKR); Knee kinematics; Ligament balance; Bellemans; Soft-tissue balance
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Prospective, single-group, non-blind, interventional study
Masking Description: Non-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single interventional group at Bærum Hopsital Vestre Viken Hospital Trust (Experimental): Patients that need ligament balancing will receive the procedure using a novel instrument under knee arthroplasty surgery. BrainLab navigation will be used to evaluate ligament balancing. Performed av Bærum Hospital Vestre Viken Hospital Trust
  Interventions: Device: A novel instrument for ligament balancing in total knee arthroplasty
- Single interventional group at OUH Ullevål Hospital (Experimental): Singel group non-blin interventional study group receiving ligament balancing performed using a novel instrument. Ligament balancing will be evaluated using conventional instruments.
  Interventions: Device: Novel Instrument for ligament balancing in knee arthroplasty

INTERVENTIONS:
Device: A novel instrument for ligament balancing in total knee arthroplasty — Patients will be evaluated perioperatively for ligament balance. When indicated, the novel instrument will guide puncturing of the medial collateral ligament in a systematic and step-wise fashion. Achieved ligament balance will be observed and controlled by computer navigation and a ligament tensor. Performed at Bærum Hospital vestre Viken Hospital Trust.
  Arms: Single interventional group at Bærum Hopsital Vestre Viken Hospital Trust
Device: Novel Instrument for ligament balancing in knee arthroplasty — Patients will be evaluated perioperatively for ligament balance. When indicated, the novel instrument will guide puncturing of the medial collateral ligament in a systematic and step-wise fashion. Achieved ligament balance will be observed and controlled by conventional methods using spatulas.
  Arms: Single interventional group at OUH Ullevål Hospital

SUMMARY:
The goal of this interventional pilot study is to evaluate if performing ligament balancing on the medial collateral ligament (MCL) in a more systematical manner with a novel instrument can produce more objective and repeatable ligament lengthening in Total Knee Arthroplasty. The main questions it aim to answer are:

1. Is it feasible to perform systematic ligament balancing on the MCL using a novel instrument?
2. Can a novel instrument for ligament balancing acquire more objective and repeatable results, without risk of injury?

Participants must consent prior to the surgery, but inclusion is only done once ligament balancing is indicated during surgery. Patients will be follow-up as standard protocol for Total Knee Arthroplasty patients at the hospital.

DETAILED DESCRIPTION:
Varus deformity is the most common deformity (60-80%) in patients undergoing total knee arthroplasty (TKA). In varus knees, there could be shortening of medial structures; therefore, if mechanical alignment is the goal, perpendicular bone cuts could produce a trapezoidal gap between the femur and tibia, with a shorter medial side. This imbalance should be corrected through ligament balancing as it is seen as a prerequisite for good function and survival. Aunan et al. found ligament balancing to be necessary in 70 of 100 consecutive TKAs.

Several ligament balancing techniques exist and most focus on lengthening the soft tissue on the concave side of the knee. Bellemans' and Whiteside's techniques are examples of ligament balancing procedures. In varus knees Bellemans' technique is performed with multiple perforations (pie-crusting) of the medial collateral ligament (MCL), while Whiteside's technique is performed with sequential ligament and soft tissue release, where the MCL is evaluated first. However, no technique has proved clinically superior to others. In traditional methods, it is difficult to reliably predict ligament lengthening and it relies on the performing surgeons' feel and experience. Aunan et al. found wide variation in lengthening achieved using Whiteside's technique. Therefore, the investigators have developed a novel device, which aspires to further develop Bellemans' technique and produce repeatable soft tissue lengthening of the MCL.

In varus knees the most important structure in ligament balancing is the superficial and deep MCL (hereafter MCL). Bellemans' technique is a proven technique, which uses an end-cutting cannula to puncture the MCL by freehand, with the objective of severing some ligament fibers. When the force applied to the ligament is kept constant, each remaining fiber will be exposed to a higher force and lengthen. Bellemans' technique lacks an objective method of guiding the puncturing, and the execution and results therefore vary. The novel instrument invented by the investigators, has a specific grid that objectively guides perpendicular puncturing using an end-cutting cannula and evenly distributes punctures throughout the ligament, which will produce a predefined spread of punctures and severing of fibers. The investigators believe this grid is key to achieving repeatable lengthening of the MCL, and promising results have been shown in porcine and human cadaveric tissue.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 40 years of age that require total knee arthroplasty
* Idiopathic osteoarthrosis, osteonecrosis or avascular osteonecrosis
* Otherwise fairly healthy/ no significant health issues

Exclusion Criteria:

* Age under 40 years of age
* Pregnant
* Revisions or reoperations
* Considerable earlier injury to the knee
* Isolated patellofemoral osteoarthrosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Is it feasible to perform systematic ligament balancing on the MCL using a novel instrument? | 1 year
  The investigators will be studying if it is possible to perform systematic ligament balancing on the MCL during total knee arthroplasty surgery, using a novel instrument.
MCL-lengthening in millimeters after ligament balancing using the novel instrument | 1 year
  The investigators will be evaluating the amount of lengthening of the medial collateral ligament (MCL) in millimeters, that is achieved when using a novel instrument for systematic ligament balancing in total knee arthroplasty. Lengthening in millimeters is evaluated using computer navigated orthopaedic surgery (CAOS) and ligament tensioners or spatulas. The investigators will evaluate if the lengthening is linear and repeatable between individuals using regression analysis.

SECONDARY OUTCOMES:
Demographic information - height (cm) - and how this parameters affects ligament balancing. | 1 year
  The investigators will evaluate if height in centimeters plays a role in how much ligament lengthening is achieved when using a novel instrument for systematic ligament balancing in MCL-lengthening. Evaluations will be done using regression analysis.
Demographic information - weight (kg) - and how this parameters affects ligament balancing. | 1 year
  The investigators will evaluate if weight in kilograms plays a role in how much ligament lengthening is achieved when using a novel instrument for systematic ligament balancing in MCL-lengthening. Evaluations will be done using regression analysis.
Demographic information - age (years) - and how this parameters affects ligament balancing. | 1 year
  The investigators will evaluate if age in years plays a role in how much ligament lengthening is achieved when using a novel instrument for systematic ligament balancing in MCL-lengthening. Evaluations will be done using regression analysis.
Demographic information - sex (biologic, male/ female) - and how this parameters affects ligament balancing. | 1 year
  The investigators will evaluate if biological sex, defined as male or female, plays a role in how much ligament lengthening is achieved when using a novel instrument for systematic ligament balancing in MCL-lengthening. Evaluations will be done using regression analysis.
Demographic information - co-morbidities (disease state) - and how this parameters affect ligament balancing. | 1 year
  The investigators will evaluate if co-morbidities, defined as disease states (eg. heart-failure, chronic lung disease, rheumatoid arthritis, etc) plays a role in how much ligament lengthening is achieved when using a novel instrument for systematic ligament balancing in MCL-lengthening. Evaluations will be done using regression analysis.
Patient reported outcome measures (PROM) using EQ-5D-5L | 1 year
  Standard protocol after total knee arthroplasty surgery at Baerum Hospital will be followed. It is standard practice to evaluate the patient health using self-assessement questionnaires at approximately 6 months. One of these questionnaires is called: EQ-5D-5L or EuroQol-5 dimension-5 Level questionnaire. It consists of 5 equally weighted dimensions with 5 equally weighted levels. The five dimensions that the questionnaire evaluates is divided into five levels of perceived problems (1-5). 1 indicates no problems and 5 indicates extreme problems. A higher level indicates more problems. The levels are combined in a 5-digit state. The minimum value is 11111 and the maximum values 55555. The combination of levels in the state indicates the severity of problems for the patient.
Patient reported outcome measures (PROM) using FJS-12 | 1 year
  Standard protocol after total knee arthroplasty surgery at Baerum Hospital will be followed. It is standard practice to evaluate the patients health using self-assessement questionnaires at approximately 6 months. One of these questionnaires is called: FJS-12 or Forgotten Joint Score 12 questions, is is designed to be used to asses artificial prosthesis awareness during daily activities following arthroplasty. The version for the knee will be used. It consists of 12 equally weighted questions that are answered on a five-level Likert scale from "never" to "mostly". Answers to each question are individually scored and summed to create a score (0-100). A low score indicates that the patient is very aware of their artificial joint and a high score indicates that the patients are very satisfied because the joint does not feel artificial.
Patient reported outcome measures (PROM) using KOOS | 1 year
  Standard protocol for Bærum Hospital and the Norwegian Registry after total knee arthroplasty surgery will be followed.One of these questionnaires is called: KOOS. KOOS is the of the most used PROMs for evaluation conditions surrounding total knee arthroplasty. KOOS-12 contains 12 items (questions). Each question is scored from 0-4, with 0 indicating no problems and 4 extreme problem. However, an overall impact score is calculated (0-100) using the 12 questions, where 0 indicates the most problematic knee and 100 the best outcome.
Coronal plane angles | 1 year
  The investigators will be evaluating the amount of lengthening of the medial collateral ligament (MCL) in millimeters, that is achieved when using a novel instrument for systematic ligament balancing in total knee arthroplasty. Lengthening in millimeters is evaluated using computer navigated orthopaedic surgery (CAOS) and ligament tensioners or spatulas. The investigators will evaluate if the lengthening is linear and repeatable between individuals using regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Lars HW Engseth, MD, Principal Investigator — Oslo University Hospital, Ullevaal, Oslo, Norway; Jarle Vik, MD, Principal Investigator — Baerum Hospital, Vestre Viken Hospital Trust, Baerum, Norway
Locations (2):
- Norway (2):
  - Bærum Hospital, Vestre Viken Hospital Trust, Bærums verk, Akershus
  - Oslo University Hospital, Ullevaal, Oslo, Oslo County

IPD SHARING:
Plan to Share IPD: No
No, due to national data protection laws.

REFERENCES:
- [Background] Verdonk PC, Pernin J, Pinaroli A, Ait Si Selmi T, Neyret P. Soft tissue balancing in varus total knee arthroplasty: an algorithmic approach. Knee Surg Sports Traumatol Arthrosc. 2009 Jun;17(6):660-6. doi: 10.1007/s00167-009-0755-7. Epub 2009 Mar 17. PMID 19290507
- [Background] Bellemans J. Multiple needle puncturing: balancing the varus knee. Orthopedics. 2011 Sep 9;34(9):e510-2. doi: 10.3928/01477447-20110714-48. PMID 21902147
- [Background] Bellemans J, Vandenneucker H, Van Lauwe J, Victor J. A new surgical technique for medial collateral ligament balancing: multiple needle puncturing. J Arthroplasty. 2010 Oct;25(7):1151-6. doi: 10.1016/j.arth.2010.03.007. Epub 2010 May 10. PMID 20452181
- [Background] Aunan E, Kibsgard T, Clarke-Jenssen J, Rohrl SM. A new method to measure ligament balancing in total knee arthroplasty: laxity measurements in 100 knees. Arch Orthop Trauma Surg. 2012 Aug;132(8):1173-81. doi: 10.1007/s00402-012-1536-1. Epub 2012 May 13. PMID 22581351
- [Background] Neogi T. The epidemiology and impact of pain in osteoarthritis. Osteoarthritis Cartilage. 2013 Sep;21(9):1145-53. doi: 10.1016/j.joca.2013.03.018. PMID 23973124
- [Background] Beswick AD, Wylde V, Gooberman-Hill R, Blom A, Dieppe P. What proportion of patients report long-term pain after total hip or knee replacement for osteoarthritis? A systematic review of prospective studies in unselected patients. BMJ Open. 2012 Feb 22;2(1):e000435. doi: 10.1136/bmjopen-2011-000435. Print 2012. PMID 22357571
- [Background] Aunan E, Rohrl SM. No detrimental effect of ligament balancing on functional outcome after total knee arthroplasty: a prospective cohort study on 129 mechanically aligned knees with 3 years' follow-up. Acta Orthop. 2018 Oct;89(5):548-554. doi: 10.1080/17453674.2018.1485283. Epub 2018 Jun 8. PMID 29883259
- [Background] Whiteside LA. Soft tissue balancing: the knee. J Arthroplasty. 2002 Jun;17(4 Suppl 1):23-7. doi: 10.1054/arth.2002.33264. PMID 12068398
- [Background] Fang DM, Ritter MA, Davis KE. Coronal alignment in total knee arthroplasty: just how important is it? J Arthroplasty. 2009 Sep;24(6 Suppl):39-43. doi: 10.1016/j.arth.2009.04.034. Epub 2009 Jun 24. PMID 19553073
- [Background] Abdel MP, Ollivier M, Parratte S, Trousdale RT, Berry DJ, Pagnano MW. Effect of Postoperative Mechanical Axis Alignment on Survival and Functional Outcomes of Modern Total Knee Arthroplasties with Cement: A Concise Follow-up at 20 Years. J Bone Joint Surg Am. 2018 Mar 21;100(6):472-478. doi: 10.2106/JBJS.16.01587. PMID 29557863
- [Background] Magnussen RA, Weppe F, Demey G, Servien E, Lustig S. Residual varus alignment does not compromise results of TKAs in patients with preoperative varus. Clin Orthop Relat Res. 2011 Dec;469(12):3443-50. doi: 10.1007/s11999-011-1988-6. Epub 2011 Jul 26. PMID 21789710
- [Background] Babazadeh S, Stoney JD, Lim K, Choong PF. The relevance of ligament balancing in total knee arthroplasty: how important is it? A systematic review of the literature. Orthop Rev (Pavia). 2009 Oct 10;1(2):e26. doi: 10.4081/or.2009.e26. PMID 21808688
- [Background] Mihalko WM, Whiteside LA, Krackow KA. Comparison of ligament-balancing techniques during total knee arthroplasty. J Bone Joint Surg Am. 2003;85-A Suppl 4:132-5. doi: 10.2106/00004623-200300004-00018. No abstract available. PMID 14652405
- [Background] Robinson JR, Bull AM, Amis AA. Structural properties of the medial collateral ligament complex of the human knee. J Biomech. 2005 May;38(5):1067-74. doi: 10.1016/j.jbiomech.2004.05.034. PMID 15797588
- [Background] Koh IJ, Kwak DS, Kim TK, Park IJ, In Y. How effective is multiple needle puncturing for medial soft tissue balancing during total knee arthroplasty? A cadaveric study. J Arthroplasty. 2014 Dec;29(12):2478-83. doi: 10.1016/j.arth.2013.11.004. Epub 2013 Nov 9. PMID 24360488
- [Background] Engseth LHW, Gronsund J, Aunan E, Brattgjerd JE, Schulz A, Moatshe G, Rohrl SM. A novel instrument for ligament balancing: a biomechanical study in human cadaveric knees. J Exp Orthop. 2023 Aug 16;10(1):83. doi: 10.1186/s40634-023-00643-7. PMID 37584812
- [Background] Liu F, Yue B, Gadikota HR, Kozanek M, Liu W, Gill TJ, Rubash HE, Li G. Morphology of the medial collateral ligament of the knee. J Orthop Surg Res. 2010 Sep 16;5:69. doi: 10.1186/1749-799X-5-69. PMID 20846377
- [Background] Aglietti P, Lup D, Cuomo P, Baldini A, De Luca L. Total knee arthroplasty using a pie-crusting technique for valgus deformity. Clin Orthop Relat Res. 2007 Nov;464:73-7. doi: 10.1097/BLO.0b013e3181591c48. PMID 17975373
- See also: National Joint Registry — https://reports.njrcentre.org.uk
- See also: The American Joint Replacement Registry Annual Report. American Academy of Orthopaedic Surgeons. — https://www.aaos.org/registries/publications/ajrr-annual-report/